CLINICAL TRIAL: NCT03477279
Title: Developing and Assessing a Male Engagement Intervention in Option B+ in Malawi: A Randomized Controlled Trial in Lilongwe
Brief Title: Developing and Assessing a Male Engagement Intervention in Option B+ in Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-0681; R00MH104154 (NIH)
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-03

CONDITIONS: Hiv
Keywords: couple HIV testing and counseling; disclosure; Malawi
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Counseling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individual (SOC) (No Intervention): HIV-infected pregnant women enrolled in the individual arm of the study will receive Standard of Care Option B+ procedures.
- Couple (Intervention) (Experimental): In addition to receiving standard of care procedures, HIV-infected pregnant women in the couple arm will be provided with an intervention aimed at recruiting their male partners, providing enhanced couple counseling and testing, engaging their male partners in their care, and supporting male partners to receive care and treatment services.
  Interventions: Behavioral: Enhanced Couple HIV Testing and Counseling
- HIV-Uninfected Cohort (No Intervention): HIV-uninfected pregnant women will be invited to participate in a cross-sectional study. No intervention will be provided and no follow-up will be conducted.

INTERVENTIONS:
Behavioral: Enhanced Couple HIV Testing and Counseling — Participants are provided study-specific partner referral cards and encouraged to bring male partners to antenatal care for a male engagement intervention. Those who do not present on their own are then traced.
  Couples will receive three enhanced couple counseling sessions that include: pre-test counseling, return of joint results, and post-test counseling. HIV-infected men will be able to initiate cART at the antenatal clinic and the couple will be offered condoms from the HTC counselor. Between sessions, couple members can pick up condoms and cART for one another.
  Other Names: male engagement intervention
  Arms: Couple (Intervention)

SUMMARY:
There is promising evidence that couple-based approaches within Malawi's Option B+ prevention of mother to child transmission program could address help address 1) poor male engagement in the HIV continuum of care, 2) low male adoption of biomedical HIV prevention approaches, 3) sub-optimal female engagement in the continuum of care, and 4) poor or uncertain infant outcomes. Our team has developed an intervention to address these challenges, and will conduct a randomized controlled trial (N=500 couples) to assess intervention effectiveness at one year. Women with recent HIV infections enrolled in this trial will be compared against a cohort of 350 HIV-uninfected women to explore predictors of HIV acquisition in pregnancy in Malawi.

DETAILED DESCRIPTION:
In sub-Saharan Africa, engaging HIV-infected men in HIV care and treatment and engaging HIV-uninfected men in prevention has proven challenging. Along all steps of the HIV care-seeking cascade, men exhibit worse care-seeking behaviors. They are less likely to seek HIV testing and counseling (HTC), initiate combination antiretroviral therapy (cART), and be retained in cART care. Poor care-seeking has resulted in a lower prevalence of viral suppression and earlier mortality. Additionally, men rarely engage in the antenatal care-seeking of their female sexual partners, leading to worse maternal and infant outcomes. This low level of engagement has been noted in Malawi's Option B+ prevention of mother to child transmission (PMTCT) program, and has been a critical barrier to female Option B+ uptake and retention, and a missed opportunity for engaging men.

There is promising evidence that couple-based approaches within Malawi's Option B+ prevention of mother to child transmission program could address all of these challenges: poor male engagement in the HIV continuum of care, low male adoption of biomedical HIV prevention approaches, sub-optimal female engagement in the continuum of care, and poor or uncertain infant outcomes. Our team has designed a couples-based intervention to address these challenges, and will conduct a randomized controlled trial (N=500 couples) to assess intervention effectiveness at one year. Results from this study are expected to inform how best to address family outcomes in an Option B+ program.

This study has the following aims described below:

Aim 1: Determine whether the couple-based intervention increases new HIV-positive diagnoses among HIV-infected male sex partners, helps HIV-infected men engage and remain in care, and contributes to male viral suppression compared to individual standard of care. The investigators will compare the couple-based intervention to standard of care for increasing the proportion of men who are aware of being HIV-infected, the proportion of these men who initiate and remain in cART care, and the proportion of these men with viral suppression at one year.

Aim 2: Determine whether the couple-based intervention identifies HIV-discordant couples and decreases the likelihood of male exposure to HIV compared to individual standard of care. The investigators will compare the intervention to standard of care for increasing the number of men with non-HIV exposure from their female partner through consistent condom use, viral suppression, abstinence, or a combination of these methods over one year.

Aim 3: Determine whether the couple-based intervention improves female cART retention and viral suppression compared to individual standard of care. The investigators will compare the intervention to standard of care for female cART retention and viral suppression at one year.

Aim 4: Determine whether the couple-based intervention improves infant early infant diagnosis uptake compared to individual standard of care. Explore uptake of early infant diagnosis and rates of mother-to-child transmission and child survival in the two intervention arms.

Aim 5: Develop an in-depth understanding of HIV transmission dynamics in Lilongwe. Using the biomarkers and behavioral survey, we will seek to understand transmission timing, direction, and context in Lilongwe. We will compare women with recent HIV infection to a population of HIV-uninfected controls (n=350) to understand predictors of HIV acquisition in pregnancy in Malawi.

ELIGIBILITY:
Inclusion Criteria (HIV-infected Women):

* HIV-infected and eligible for Option B+
* >18 years old or 15-17 years old and married
* Planning to remain in the Bwaila catchment area for the next year or notify the study team if they leave the area or change facilities
* Part of a heterosexual relationship for >3 months

  * Expects the partner to be in the relevant catchment area for at least one week in the next six months.
  * Able and willing to give locator information for this partner
  * Willing to have study staff conduct phone and physical tracing of that partner
  * Willing to undergo a couple-based intervention with this partner
* Able and willing to provide informed consent

Inclusion Criteria (Male Partners of HIV-infected women)

* >18 years old or 15-17 years old and married
* In a relationship with the female partner for >3 months

  * Willing to undergo a couples-based intervention with their female partner
* Able and willing to provide informed consent

Inclusion Criteria (HIV-uninfected Women):

* HIV-uninfected
* >18 years old or 15-17 years old and married
* Part of a heterosexual relationship for >3 months

  * Expects the partner to be in the relevant catchment area for at least one week in the next six months.
  * Willing to receive couples-based HIV testing and counseling with this partner
* Able and willing to provide informed consent

Exclusion Criteria (all Women and Male Partners):

• Any condition that in the opinion of the study investigator would compromise the ability of the prospective participant to provide informed consent, undergo study procedures safely, or would prevent proper conduct of the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nora E Rosenberg, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Bwaila District Hospital Antenatal Unit, Lilongwe, Central District, Malawi

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Individual (HIV+ Women): HIV-infected pregnant women enrolled in the individual arm of the study will receive Standard of Care Option B+ procedures.
- Couple (HIV+ Women): These women will receive 1) support to recruit their male partners, 2) enhanced couple counseling and testing, and 3) support for male partner engagement in care.
- Male Partners of Women in Individual: These men will have access to standard of care procedures.
- Male Partners of Women in Couple: These men will receive 1) support with recruitment, 2) enhanced couple counseling and testing, and 3) support for engagement in care.
- Control Population (HIV- Women): HIV-negative pregnant women will be invited to participate in a cross-sectional study. No intervention will be provided and no follow-up will be conducted.
Period: Overall Study
Arm/Group | Individual (HIV+ Women) | Couple (HIV+ Women) | Male Partners of Women in Individual | Male Partners of Women in Couple | Control Population (HIV- Women)
Started | 250 | 250 | 98 | 168 | 350
Completed | 203 | 202 | 98 | 136 | 349
Not Completed | 47 | 48 | 0 | 32 | 1

BASELINE CHARACTERISTICS:
Population: Data unreported for 6 surveys that corrupted during upload. Data unavailable for one HIV-negative woman.
Groups:
- Individual (HIV+ Women): HIV-positive pregnant women enrolled in the Individual arm will receive Standard of Care Option B+ procedures.
- Couple (HIV+ Women): HIV-positive pregnant women enrolled in the Couple arm will receive 1) support to recruit their male partners, 2) enhanced couple counseling and testing, and 3) support for male partner engagement in care.
- Total: Total of all reporting groups
Arm/Group | Individual (HIV+ Women) | Couple (HIV+ Women) | Male Partners of Women in Individual | Male Partners of Women in Couple | Control Population (HIV- Women) | Total
Number analyzed (Participants) | 246 | 249 | 98 | 167 | 349 | 1109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 11 | 1 | 0 | 37 | 64
  Between 18 and 65 years | 231 | 238 | 97 | 167 | 312 | 1045
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246 | 249 | 0 | 0 | 349 | 844
  Male | 0 | 0 | 98 | 167 | 0 | 265
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 246 | 249 | 98 | 167 | 349 | 1109

OUTCOME MEASURES:

1. Primary Outcome: Number of Women Retained in Care
Description: Women who presented at 12 months and reported taking at least one dose of ART in the last seven days
Time Frame: 12 months
Population: This is an HIV-positive female only outcome. 134 HIV-positive women did not present for the 12 month study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Individual (HIV+ Women) | Couple (HIV+ Women)
Number analyzed (Participants) | 181 | 185
Participants | 160 | 164
Statistical Analysis 1: Comparison: Individual (HIV+ Women) vs Couple (HIV+ Women); Test type: Superiority; Risk Difference (RD) = 0.9, 95% CI 2-sided [-5.6 to 7.3] — Couple (HIV+ Women) - Individual (HIV+ Women)

2. Primary Outcome: Number of Women With Viral Suppression
Description: Women who presented at 12 months with a viral load <1000 copies/mL
Time Frame: 12 months
Population: This is an HIV-positive female only outcome.138 HIV-positive women did not present for the 12 month study visit or did not provide the blood sample required for viral load ascertainment
Measure: Count of Participants; unit: Participants
Arm/Group | Individual (HIV+ Women) | Couple (HIV+ Women)
Number analyzed (Participants) | 178 | 184
Participants | 145 | 162
Statistical Analysis 1: Comparison: Individual (HIV+ Women) vs Couple (HIV+ Women); Test type: Superiority; Risk Difference (RD) = 6.6, 95% CI 2-sided [-0.8 to 14.0] — Couple (HIV+ Women) - Individual (HIV+ Women)

3. Primary Outcome: Number of HIV-positive Male Partners Aware of Their HIV-positive Status
Description: HIV-positive male partners who presented at 12 months and reported knowing they were HIV-positive prior to receiving the results of the HIV test conducted at the 12 month study visit
Time Frame: 12 months
Population: This is a male only outcome. 141 men did not present at 12 months, or refused HIV testing at 12 months, or tested HIV-negative/indeterminate at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Male Partners of Women in Individual | Male Partners of Women in Couple
Number analyzed (Participants) | 53 | 72
Participants | 44 | 67
Statistical Analysis 1: Comparison: Male Partners of Women in Individual vs Male Partners of Women in Couple; Test type: Superiority; Risk Difference (RD) = 10.0, 95% CI 2-sided [-1.7 to 21.7] — Male Partners of Women in Couple - Male Partners of Women in Individual

4. Primary Outcome: Number of HIV-positive Male Partners Retained in Care
Description: HIV-positive male partners who presented at 12 months and reported taking at least one dose of ART in the last seven days
Time Frame: 12 months
Population: This is a male only outcome. 142 men did not present at 12 months, or refused HIV testing at 12 months, or tested HIV-negative/indeterminate at 12 months, or did not report information on ART use
Measure: Count of Participants; unit: Participants
Arm/Group | Male Partners of Women in Individual | Male Partners of Women in Couple
Number analyzed (Participants) | 52 | 72
Participants | 34 | 59
Statistical Analysis 1: Comparison: Male Partners of Women in Individual vs Male Partners of Women in Couple; Test type: Superiority; Risk Difference (RD) = 16.6, 95% CI 2-sided [0.9 to 32.3] — Male Partners of Women in Couple - Male Partners of Women in Individual

5. Primary Outcome: Number of HIV-positive Male Partners With Viral Suppression
Description: HIV-positive male partners who presented at 12 months with a viral load <1000 copies/mL
Time Frame: 12 months
Population: This is a male only outcome. 141 men did not present at 12 months, or refused HIV testing at 12 months, or tested HIV-negative/indeterminate at 12 months, or did not provide the blood sample required for viral load ascertainment
Measure: Count of Participants; unit: Participants
Arm/Group | Male Partners of Women in Individual | Male Partners of Women in Couple
Number analyzed (Participants) | 53 | 72
Participants | 31 | 53
Statistical Analysis 1: Comparison: Male Partners of Women in Individual vs Male Partners of Women in Couple; Test type: Superiority; Risk Difference (RD) = 15.1, 95% CI 2-sided [-1.6 to 31.8]

6. Primary Outcome: Number of HIV-negative Men Without HIV Exposure From Their Primary Partner
Description: HIV-negative men with a) consistent condom use in the last six months or b) a suppressed female partner or c) abstinence with primary partner
Time Frame: 12 months
Population: This is a male only outcome. 162 did not present at 12 months, or refused HIV testing at 12 months, or tested HIV-positive/indeterminate at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Male Partners of Women in Individual | Male Partners of Women in Couple
Number analyzed (Participants) | 41 | 63
Participants | 39 | 59
Statistical Analysis 1: Comparison: Male Partners of Women in Individual vs Male Partners of Women in Couple; Test type: Superiority; Risk Difference (RD) = -2.4, 95% CI 2-sided [-13.2 to 8.5] — Male Partners of Women in Couple - Male Partners of Women in Individual

7. Secondary Outcome: Number of HIV-positive Female Participants Who Reported Early Infant Diagnosis
Description: HIV-positive female participants who reported a live birth and uptake of early infant diagnosis
Time Frame: 12 months
Population: This is an HIV-positive female only outcome. For 154 observations, there was no data available on infant outcomes or no live birth
Measure: Count of Participants; unit: Participants
Arm/Group | Individual (HIV+ Women) | Couple (HIV+ Women)
Number analyzed (Participants) | 171 | 175
Participants | 162 | 158
Statistical Analysis 1: Comparison: Individual (HIV+ Women) vs Couple (HIV+ Women); Test type: Superiority; Risk Difference (RD) = -4.5, 95% CI 2-sided [-10.0 to 10.7] — Couple (HIV+ Women) - Individual (HIV+ Women)

8. Secondary Outcome: Predictors of Recent HIV Infection
Description: Risk factor analysis to identify predictors of recent HIV infection among pregnant women
Time Frame: At the day of female consent
Population: This is a female only outcome. Of the 500 HIV-positive women enrolled into the study, 44 were classified as having recently acquired HIV. Data unavailable for one HIV-negative woman.
Measure: Count of Participants; unit: Participants
Groups:
- Individual and Couple HIV-positive Women: A subset of HIV-positive pregnant women enrolled in the individual arm and couple arms of the study with recently acquired HIV infection
Arm/Group | Individual and Couple HIV-positive Women | Control Population (HIV- Women)
Number analyzed (Participants) | 44 | 349
Participants
  Married to Primary Partner | 38 | 338
  Not Married to Primary Partner | 6 | 11
Statistical Analysis 1: Comparison: Individual and Couple HIV-positive Women vs Control Population (HIV- Women); Test type: Other; Odds Ratio (OR) = 4.9, 95% CI 2-sided [1.7 to 13.9]

ADVERSE EVENTS:
Time Frame: For the two groups of HIV-positive women, adverse event data were collected from the signing of the Informed Consent through 1 year afterward. For the two groups of male partners of HIV-positive women, adverse event data were collected from the signing of the Informed Consent through 1 year after consent of their partner.
Description: Participants in the Control arm did not receive the study intervention; therefore, adverse event information was not collected.
Arm/Group | Individual (HIV+ Women) | Couple (HIV+ Women) | Male Partners of Women in Individual | Male Partners of Women in Couple | Control Population (HIV- Women)
All-Cause Mortality (participants affected / at risk) | 1/250 | 1/250 | 0/98 | 0/168 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/250 | 0/250 | 0/98 | 0/168 | 0/0
Other Adverse Events (participants affected / at risk) | 0/250 | 0/250 | 0/98 | 0/168 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT03477279/Prot_SAP_000.pdf